CLINICAL TRIAL: NCT01282034
Title: Multicenter Randomized Controlled Trial for the Treatment of Knee Chondral and Osteochondral Lesions: Marrow Stimulation Techniques vs MaioRegen
Brief Title: Study for the Treatment of Knee Chondral and Osteochondral Lesions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fin-Ceramica Faenza Spa (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ORT-12
Record Dates: First submitted 2011-01-21; First posted 2011-01-24 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Knee Chondral Lesion; Knee Osteochondral Lesion
Keywords: CHONDRAL; OSTEOCHONDRAL
MeSH Terms: interventions — Arthroplasty, Subchondral

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Marrow stimulation (Active Comparator)
  Interventions: Procedure: Marrow stimulation - Drilling or Microfractures
- Medical device: MaioRegen (Experimental)
  Interventions: Device: MaioRegen Surgery

INTERVENTIONS:
Procedure: Marrow stimulation - Drilling or Microfractures — Subchondral drilling consists in penetration of the subchondral bone endplate and creation of holes, and it is mostly indicated for the treatment of osteochodral lesion.
  Microfractures (MF), according to Steadman's technique, are one of the most used first-line treatment for cartilage injuries, and commonly considered safe and effective.
  Other Names: subchondral Drilling; Steadman's Microfractures
  Arms: Marrow stimulation
Device: MaioRegen Surgery — MaioRegen® (is a bioceramic, multi-layered scaffold, in a single gradient structure, consisting of deantigenated Type I equine collagen and Magnesium enriched-Hydroxyapatite, able to mime the entire osteocartilaginous section. MaioRegen® is able to promote the tissue regeneration in case of severe and large chondral/osteochondral lesions.
  Other Names: osteochondral scaffold
  Arms: Medical device: MaioRegen

SUMMARY:
INTRODUCTION Marrow stimulation techniques as subchondral drilling or microfractures represent ones of the most frequently used methods for chondral and osteochodral defects repair and considered as standard techniques.

MaioRegen® (Fin-Ceramica Faenza S.p.A., Italy) is a bioceramic, multi-layered scaffold, in a single gradient structure, consisting of deantigenated Type I equine collagen and Magnesium enriched-Hydroxyapatite, able to mime the entire osteocartilaginous section. MaioRegen® is able to promote the tissue regeneration in case of severe and large chondral/osteochondral lesions, otherwise difficult to treat, as previously demonstrated in vitro, in vivo and in a clinical study.

OBJECTIVES The present study proposes to compare MaioRegen® performances with respect to reference standard surgical techniques (microfractures and subchondral drilling) for the treatment of chondral/osteochondral lesions, in order to consolidate MaioRegen®, as innovative surgical approach.

STUDY DESIGN The clinical trial is multicenter, prospective, randomized, controlled, two-arm, single-blind and involves eleven European centres and 150 patients. Eligible subjects will be randomly allocated to one of the two treatment groups: control group, treated with marrow stimulation techniques, and treatment group, treated with MaioRegen® implant.

Patient defect will be evaluated pre-operatively and each patient enrolled must meet all the entry criteria for the trial. Before enrolment, each subject should declare his voluntary participation to the study by informed consent signature.

Arthroscopic control will be carried out immediately before the randomization and thus surgical treatment, to confirm the characteristics of the lesion to be treated and finalizing the recruitment.

For each patient 6, 12 and 24 months post-operative follow-up visits will be carried out and during each follow-up visit the Case Report Form (CRF) will be filled in the specific section.

Within the CRF, at each follow-up section, commonly used and specific scores will be assigned for the established end-points (IKDC, KOOS, Tegner Score, VAS, MRI Mocart Scoring System).

Patients selected will be randomized to undergo one of two study groups, as prescribed by the randomization list.

DETAILED DESCRIPTION:
Post-operative MRI exams will be carried out for each patient during the follow-up visit, at 6, 12 and 24 months post-op., and centrally blind evaluated by two senior radiologists.

STATISTICS The study has been designed to demonstrate the superiority of MaioRegen® compared to marrow stimulation techniques.

On the basis of previous evidence and, assuming a minimum difference in the modification of the IKDC Subjective Knee Evaluation Score between MaioRegen® and the control therapy, the sample size was estimated in 74 patients for group (power=90%, first type error α=5%, drop-outs=10%), for a total sample size of 148 subjects.

The analysis of the primary end-point will be the evaluation of change from baseline to two years, in IKDC Subjective Knee Evaluation Score, comparing the results between the two groups.

Secondary end-points (functional improvement, quality of life improvement, tissue regeneration) will undergo the same analyses as the primary end-point, for each follow-up visit.

Frequency tables will be provided for overall judgement of the treatment. The incidence and gravity frequency of eventual events after surgery will be tabulated.

The study will be conducted after approval by the ethics committee board of each centre and possibly by the national competent authorities.

ELIGIBILITY:
Inclusion Criteria:

1. Patients provided written informed consent;
2. Patients aged between 18 and 60 years;
3. Knee symptomatic chondral lesion of grade III/IV (according to Outerbridge Classification) or osteochondral lesion;
4. Not re-fixable OCD lesions;
5. Lesion between 2-9 cm2;
6. Single lesion;
7. Patients agreed to actively participate in the rehabilitation protocol and follow-up program;
8. Male or female patients;
9. Women of childbearing age had to use a proven method to prevent pregnancy, before the surgical treatment.

Exclusion Criteria:

1. Patients incapable to understanding and will;
2. Patients participating in previous, concurrent or not, trials (ongoing or completed within 3 months);
3. Patients surgically treated for the same defect within one year;
4. Known allergy to collagen or calcium-phosphates;
5. Patients affected by malignancy;
6. Patients affected by metabolic or thyroid disorders;
7. Patients used to alcohol or drug (medication) abuse;
8. Patients affected by advanced osteoarthritis (Kellgren-Lawrence grade ≥3);
9. Patients affected by synovitis;
10. Untreated patellofemoral malalignment;
11. Varus or valgus malalignment exceeding 5°;
12. Body Mass Index > 30;
13. Patients previously treated for total or partial meniscectomy (>50% of the meniscus dimension);
14. Multiple lesions;
15. Kissing lesions;
16. Chondral/osteochondral tibial plate defects;
17. Concomitant menisci and chondral/osteochondral defects to be treated;
18. Untreated knee ligament instability.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 145 (Actual)
Dates: Start 2011-01; Primary Completion 2015-09 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
IKDC Subjective Knee Evaluation Form-2000 | two years

SECONDARY OUTCOMES:
IKDC Knee Examination Form-2000 | six months and one year
KOOS | six months, one year, two years
Tegner score | six months, one year, two years
VAS (Visual Analogue Scale) for pain evaluation | six months, one year, two years
MRI exam and MOCART score | six months, one year, two years

CONTACTS AND LOCATIONS:
Overall Officials: Maurilio Marcacci, Prof., Principal Investigator — Istituti Ortopedici Rizzoli
Locations (10):
- AKH University Hospital, Vienna, Vienna, Austria
- Gent Univeristy Hospital, Ghent, Belgium
- University Medical Center, Freiburg im Breisgau, Freiburg Im Breisgau, Germany
- Italy (2):
  - Istituti Ortopedici Rizzoli, Bologna, Bologna
  - Ospedal Sacro Cuore Don Calabria, Negrar, Verona
- Oslo University Hospital HF, Oslo, Norway
- District hospital of orthopaedics, Piekary Śląskie, Katowice, Poland
- Sport Science Orthopaedic Clinic, CapeTown, South Africa
- Kungsbacka Hospital, Kungsbacka, Sweden
- Schulthess Klinik, Zurich, Canton of Zurich, Switzerland